CLINICAL TRIAL: NCT02987231
Title: Electrical Stimulation Effect on Coronally Advanced Flap for the Treatment of Gingival Recession: Randomized Controlled Clinical Trial
Brief Title: Electrical Stimulation Effect on Coronally Advanced Flap
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Mauro Pedrine Santamaria, Assistant Professor, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UEPJMF 5
Record Dates: First submitted 2016-12-06; First posted 2016-12-08 (Estimated); Results first posted 2019-08-07 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Gingival Recession, Generalized
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CAF + SHAM (Sham Comparator): CAF treatment was performed by starting with two divergent releasing incisions lateral to the recessed area. A sulcular incision was made to unite the releasing incisions and the flap was raised beyond the mucogingival junction (MGJ) in split-full-split thickness. Sling sutures were placed to stabilize the flap in a coronal position 2 mm above the CEJ, followed by interrupted sutures to close the releasing incisions. Patients randomized to the SHAM Group will receive the simulation of the electrical stimulation process.
  Interventions: Procedure: CAF; Device: SHAM
- CAF + ES (Experimental): CAF treatment was performed by starting with two divergent releasing incisions lateral to the recessed area. A sulcular incision was made to unite the releasing incisions and the flap was raised beyond the mucogingival junction (MGJ) in split-full-split thickness. Sling sutures were placed to stabilize the flap in a coronal position 2 mm above the CEJ, followed by interrupted sutures to close the releasing incisions. For electrical stimulation, a unit consisting of a signal generator, a power supply, and circuit board will be used. Conductive electrodes for electrical current application will be applied to the vestibular gingival surface on each side of the flap, at a distance of 3 mm from the relaxing incisions and an alternating current of 100 μA at 9 kHz, will be distributed in order to traverse the operated area. A single application of electrical stimulation will be given for 120 seconds, once a day for five days after surgery.
  Interventions: Procedure: CAF; Device: ES

INTERVENTIONS:
Procedure: CAF — Periodontal plastic surgery for root coverage by the trapezoidal flap
  Other Names: Periodontal plastic surgery
Device: ES — Local electric stimulation for 120 seconds, once a day for a week
  Other Names: Local electric stimulation
  Arms: CAF + ES
Device: SHAM — Simulation of electric stimulation protocol. In Sham stimulation non current will be applied
  Arms: CAF + SHAM

SUMMARY:
The objective of this study is to evaluate clinically and through the concentration of inflammatory markers, the results of 6 months of electrical stimulation associated with coronally advanced flap for treatment of gingival recession.

DETAILED DESCRIPTION:
This is a prospective, parallel and controlled clinical trial. The population evaluated in the study was selected at Institute of Science and Technology (ICT), São José dos Campos, College of Dentistry.

Sixty patients presenting gingival recession will be divided in 2 groups:

* CAF group: coronally advanced flap for root coverage and sham electrical stimulation
* CAF+ES group: coronally advanced flap for root coverage plus electrical stimulation.

All surgical procedures were performed by a single operator (MPS). The gingival recession defects were randomly treated by either the trapezoidal-type of coronally advanced flap plus connective tissue graft (CAF+CTG). In brief description, CAF treatment was performed by starting with two divergent releasing incisions lateral to the recessed area. A sulcular incision was made to unite the releasing incisions and the flap was raised beyond the mucogingival junction (MGJ) in split-full-split thickness. The connective tissue graft was removed from the palate and sutured in position. Sling sutures were placed to stabilize the flap in a coronal position 2 mm above the cement-enamel junction (CEJ), followed by interrupted sutures to close the releasing incisions.

For electrical stimulation, a unit consisting of a signal generator (WaveFactoryCo., Ltd., Tokyo, Japan), a power supply (KikusuiElectronicsCo., Ltd., Tokyo, Japan) and circuit board will be used. Conductive electrodes for electrical current application will be applied to the vestibular gingival surface on each side of the flap, at a distance of 3 mm from the relaxing incisions and an alternating current of 100 microamperes (μA) at 9 kilohertz (kHz), will be distributed in order to traverse the operated area. A single application of electrical stimulation will be given for 120 seconds, once a day for a week. The electric current will have its visualization optimized through an oscilloscope. Patients randomized to the Control Group (SHAM) will receive the simulation of the electrical stimulation (ES) process.

Clinical, esthetics, and comfort of patients parameters were assessed at 45 days, 2, 3 and 6 months after the procedure.

Quantitative data were recorded as mean ± standard deviation (SD), and normality was tested using Shapiro-Wilk tests. The probing depth (PD), relative gingival recession (RGR), clinical attachment level (CAL), keratinized tissue thickness (KTT), keratinized tissue width (KTW), and dentin hypersensitivity (DH) values were examined by two-way repeated measures ANOVA to evaluate the differences within and between groups, followed by a Tukey test for multiple comparisons when the Shapiro-Wilk p value was ≥ 0.05. Those presenting Shapiro-Wilk p values < 0.05 were analyzed using a Friedman test (for intragroup comparisons) and Mann-Whitney tests (for intergroup comparisons). Patients' esthetics and discomfort measures using visual analog scale (VAS) were analyzed by T-tests. The frequency of complete root coverage was compared using χ2 tests. Intergroup root coverage esthetic score (RES) comparisons were performed with a T-test. A significance level of 0.05 was adopted.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting Miller class I or II gingival recession in the maxillary canines or premolars
* Visible cemento-enamel junction (CEJ) with pulp vitality;
* Patients presenting no signs of active periodontal disease and full-mouth plaque and bleeding score ≤20%;
* Patients older than 18 years old; probing depth ˂3 mm in the included teeth;
* Patients who agreed to participate and signed an informed consent form.

Exclusion Criteria:

* Patients presenting systemic problems that would contraindicate the surgical procedure;
* Patients taking medications known to interfere with the wound healing process or that contraindicate the surgical procedure;
* Smokers or pregnant women;
* Patients who underwent periodontal surgery in the area of interest;
* Patients with orthodontic therapy in progress.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-11; Primary Completion 2017-09 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mauro P Santamaria, PhD, Principal Investigator — ICT-UNESP
Locations (1):
- Felipe Lucas da Silva Neves, São José dos Campos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] de Sanctis M, Zucchelli G. Coronally advanced flap: a modified surgical approach for isolated recession-type defects: three-year results. J Clin Periodontol. 2007 Mar;34(3):262-8. doi: 10.1111/j.1600-051X.2006.01039.x. PMID 17309597
- [Background] Tomofuji T, Ekuni D, Azuma T, Irie K, Endo Y, Kasuyama K, Nagayama M, Morita M. Effects of electrical stimulation on periodontal tissue remodeling in rats. J Periodontal Res. 2013 Apr;48(2):177-83. doi: 10.1111/j.1600-0765.2012.01518.x. Epub 2012 Aug 14. PMID 22891771

RESULTS

PARTICIPANT FLOW:
Recruitment Details: At clinical site
Pre-assignment Details: The study recruited 66 eligible patients. However, three patients were excluded before assignment to groups. Two recruited patients never presented for treatment and one declined to proceed.
Groups:
- CAF + ES: CAF treatment was performed by starting with two divergent releasing incisions lateral to the recessed area. The flap was raised beyond the mucogingival junction (MGJ) in split-full-split thickness. Sling sutures were placed to stabilize the flap in a coronal position 2 mm above the CEJ. For electrical stimulation, a unit consisting of a signal generator, a power supply, and a circuit board will be used. Conductive electrodes for electrical current application will be applied to the vestibular gingival surface on each side of the flap, at a distance of 3 mm from the relaxing incisions and an alternating current of 100 μA at 9 kHz, will be distributed in order to traverse the operated area. A single application of electrical stimulation will be given for 120 seconds, once a day for five days after surgery.
  CAF: Periodontal plastic surgery for root coverage by the trapezoidal flap
  ES: Local electric stimulation for 120 seconds, once a day for a week
Period: Overall Study
Arm/Group | CAF + SHAM | CAF + ES
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CAF + SHAM | CAF + ES | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 30 | 29 | 59
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (12.68) | 39.86 (10.14) | 41.13 (11.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 21 | 39
  Male | 12 | 9 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 2 | 7
  White | 24 | 28 | 52
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Brazil | 30 | 30 | 60
Gingival recession depth [Mean (Standard Deviation); unit: millimeters] | 3.09 (0.41) | 3.2 (0.58) | 3.18 (0.11)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Defect Coverage
Description: Percentage mean (%) of root surface covered by the surgical treatment, measured through a periodontal probe.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percentage of root coverage
Arm/Group | CAF + SHAM | CAF + ES
Number analyzed (Participants) | 30 | 30
percentage of root coverage | 79.47 (21.19) | 85.97 (17.41)

2. Secondary Outcome: Root Coverage Esthetic Score
Description: The Root Coverage Esthetic Scale (RES; Cairo et al. 2009) was performed by two blinded and independent examiners (CFA and IFM) at the 6-month post-operative assessment. This score evaluates five variables: level of the gingival margin, marginal tissue contour, soft tissue texture, mucogingival junction alignment, and gingival color. Because complete root coverage was the primary treatment goal, and the other variables were considered secondary, the value assigned for root coverage was 60% of the total score, whereas 40% was assigned to the other four variables. With regard to the assessment of the final position of the gingival margin, 3 points were given for partial root coverage, and 6 points were given for complete root coverage; 0 points were assigned when the final position of the gingival margin was equal or apical to the previous recession. One point was assigned for each of the other four variables. The final score ranged from 0-10, higher values were considered better.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CAF + SHAM | CAF + ES
Number analyzed (Participants) | 30 | 30
units on a scale | 8.03 (0.37) | 7.9 (0.23)

ADVERSE EVENTS:
Time Frame: The period of data collection related to adverse effects started in the immediate postoperative period up to 6 months of follow-up.
Arm/Group | CAF + SHAM | CAF + ES
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-08-15): https://cdn.clinicaltrials.gov/large-docs/31/NCT02987231/Prot_SAP_000.pdf